CLINICAL TRIAL: NCT04077268
Title: Becoming Traumatic Brain Injured Patients at Day 7 of Their Trauma in Poitiers Emergency
Brief Title: Becoming Traumatic Brain Injured Patients at Day 7 of Their Trauma
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Distance
Record Dates: First submitted 2019-05-28; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: GOS-E — Call at 7 days, patients add a brain trauma to know their sequeals

SUMMARY:
To study the future of traumatic brain injured patients at day 7 of their trauma

Primary endpoint: Fate, classified as survival with or without sequelae, death. Use of the GOS-E scale to classify survival with or without sequelae. The collection of this scale will be done by telephone contact, 7 days of admission to the emergency room.

Secondary judgment criteria:

* Compendium of the realization of the CT / time respected between the TCL and the CT / Hospitalization / 2nd CT to realize at 24 hours in the patients treated by TAC or AAP
* Application of the recommendations of the French Society of Emergency Medicine 2012: Become 7 days of patients classified according to whether or not the recommendations, .
* Become TCL patients under AAP or TAC
* Number of reconsultation, rehospitalization, new imaging within 7 days after TCL

ELIGIBILITY:
Inclusion Criteria:

* Patient of both sexes, at least 18 years old,
* Patient with mild head trauma, Glasgow 13-15
* Patient without tutorship or curatorship
* Affiliation to social security
* No opposition of the patient or relatives to participation in the study.

Exclusion Criteria:

* Patient already included in this study
* Refusal to participate in this search
* Patient undergoing enhanced protection (persons deprived of liberty by a judicial or administrative decision, adults under legal protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient add a head mild trauma and consult at the emergency of Poitiers
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Becoming of traumatic brain injured patients: becoming classified in alive with or without sequelae or death, by using scale of GOS E | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of POITIERS, Poitiers, France

IPD SHARING:
Plan to Share IPD: No